CLINICAL TRIAL: NCT06818786
Title: Effects of New Pictorial Cigarette Pack Warnings on Vietnamese Smokers' Perceptions and Smoking Behaviors: A Randomized Controlled Trial
Brief Title: Effects of New Pictorial Cigarette Pack Warnings on Vietnamese Smokers' Perceptions and Smoking Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Hanoi University of Public Health (Other)
Responsible Party: Principal Investigator, Thi Phuong Thao Tran, Principal Investigator, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H25022
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pictorial Health Warnings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Branded pack with a new set of 6 PHWs covering 50% of cigarette packs without quitline information (Experimental)
  Interventions: Other: Branded pack with new PHWs covering 50% of the pack without quitline information
- Branded pack with a new set of 6 PHWs covering 85% of cigarette packs without quitline information (Experimental)
  Interventions: Other: Branded pack with new PHWs covering 85% of the pack with quitline information
- Branded pack with a new set of 6 PHWs covering 85% of cigarette packs with quitline information (Experimental)
  Interventions: Other: Branded pack with new PHWs covering 85% of the pack without quitline information
- Plain pack with new PHWs covering 85% of the pack with quitline information (Experimental)
  Interventions: Other: Plain pack with new PHWs covering 85% of the pack with quitline information
- Branded pack with the current set of PHWs covering 50% of the pack without quitline information (Active Comparator)
  Interventions: Other: Branded pack with the current set of PHWs covering 50% of the pack without quitline information

INTERVENTIONS:
Other: Branded pack with new PHWs covering 50% of the pack without quitline information — Participants received and were required to view six images depicting a branded cigarette pack with a new set of six pictorial health warnings covering 50% of the pack, without quitline information.
  Arms: Branded pack with a new set of 6 PHWs covering 50% of cigarette packs without quitline information
Other: Branded pack with new PHWs covering 85% of the pack without quitline information — Participants received and were required to view six images depicting a branded cigarette pack with a new set of six pictorial health warnings covering 85% of the pack, without quitline information.
  Arms: Branded pack with a new set of 6 PHWs covering 85% of cigarette packs with quitline information
Other: Branded pack with new PHWs covering 85% of the pack with quitline information — Participants received and were required to view six images depicting a branded cigarette pack with a new set of six pictorial health warnings covering 85% of the pack, with quitline information
  Arms: Branded pack with a new set of 6 PHWs covering 85% of cigarette packs without quitline information
Other: Plain pack with new PHWs covering 85% of the pack with quitline information — Participants received and were required to view six images depicting a plain cigarette pack with a new set of six pictorial health warnings covering 85% of the pack, with quitline information
  Arms: Plain pack with new PHWs covering 85% of the pack with quitline information
Other: Branded pack with the current set of PHWs covering 50% of the pack without quitline information — Participants received and were required to view 6 images depicting a branded cigarette pack with a current set of 6 pictorial health warnings covering 50% of cigarette packs without quitline information (It is the current pictorial health warnings implemented in Vietnam)
  Arms: Branded pack with the current set of PHWs covering 50% of the pack without quitline information

SUMMARY:
This proposed study will assess the effects of different scenarios of PHW policies on smokers' reactions to warnings, attitudes and beliefs, behavioral intentions, and quitting behaviors, with specific aims: 1) to assess the impact of new PHWs covering 50% of cigarette packs, 2) to assess the impact of new larger PHWs covering 85% of cigarette packs, 3) to assess the impact of incorporating quitline information on cigarette packs, and 4) to assess the impact of plain packaging. These aims will be achieved by conducting a five-arm RCT among 1000 adult smokers (n=200 per arm). It includes four intervention groups: 1) branded pack with a new set of 6 PHWs covering 50% of cigarette packs without quitline information, 2) branded pack with a new set of 6 PHWs covering 85% of cigarette packs without quitline information, 3) branded pack with a new set of 6 PHWs covering 85% of cigarette packs with quitline information, and 4) plain pack with a new set of 6 PHWs covering 85% of cigarette packs with quitline information. A control group will use branded packs with the current set of 6 PHWs, covering 50% of cigarette packs without quitline information.

Given that the pictorial health warnings (PHW) on cigarette packs need to be renewed, this project will provide highly policy-relevant and timely scientific evidence on the effect of new PHW policies in Vietnam. Additionally, this project would be the first to address the research gap in understanding the effect of adding quitline information to PHWs-a gap not explored in previous studies. With the potential for significant outcomes, the findings will help Vietnamese policymakers enact stronger PHW policies in upcoming years, aiming to increase perceived harms of smoking and foster smoking cessation, ultimately saving millions of lives in Vietnam

ELIGIBILITY:
Inclusion Criteria:

* having smoked at least 100 cigarettes in their lifetime and currently smoking
* aged 18 or older
* fluent in Vietnamese
* smartphone users

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2024-08-24 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Emotional and cognitive responses | At the enrollment
  Negative emotions, including sadness, anger, fear, guilt, disgust, worry, and shame, were measured on a scale from 1 (not at all) to 9 (extremely).
  Perceived message effectiveness was assessed using the following statements:
  "This warning discourages me from wanting to smoke." "This warning makes smoking seem unpleasant to me." "This warning makes me concerned about the health effects of smoking." Participants rated their agreement on a scale from 1 (strongly disagree) to 7 (strongly agree), with an additional "don't know" option.

SECONDARY OUTCOMES:
Attitudes and beliefs | At the enrollment
  Health risk perceptions were assessed using the following questions:
  "If you were to smoke cigarettes every day, how likely is it that they would harm your overall health?" "If you were to smoke cigarettes every day, how likely is it that you would get addicted?" Participants rated their responses on a scale from 1 (not at all likely) to 5 (extremely likely), with an additional "don't know" option.
  Health-related beliefs were assessed using the following statements:
  "Tobacco smoke is dangerous for non-smokers' health." "Smoking causes lung cancer." "Smoking causes oral cancer." "Smoking causes bleeding in the brain and stroke." "Smoking causes neck cancer." Participants rated their agreement on a scale from 1 (strongly disagree) to 7 (strongly agree), with an additional "don't know" option.
Behavioral intentions | At the enrollment
  Behavioral intentions were assessed using the following questions:
  Quit motivation: "How motivated are you to quit smoking in the next month?" Quit intention: "How likely are you to quit smoking in the next month?" Quitline call intention: "How likely are you to call the quitline in the next month?" Participants rated their responses on a scale from 1 (not at all) to 9 (extremely).
Recall and behavioral outcomes at 2-week follow-up | at 2 weeks
  This study assessed various recall and behavioral outcomes at 2 -week follow-up, including whether participants had thought about the harms of smoking, recalled the national quitline number, engaged in communication behaviors related to smoking and quitting, forwent cigarettes due to harm-related thoughts, made a quit attempt, or reduced the number of cigarettes smoked per day after 2 weeks. All outcomes were recorded as binary (Yes/No).

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi University of Public Health, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided